CLINICAL TRIAL: NCT05703451
Title: Prevalence and Severity of Surgical Adhesions Among Women Undergoing Laparoscopic Surgery at Women's Health Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Shaban Mohammed Farghaly, resident doctor, Assiut University
Other Study IDs: surgical adhesions
Record Dates: First submitted 2023-01-09; First posted 2023-01-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Surgical Adhesions
MeSH Terms: conditions — Tissue Adhesions | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: laparoscopic surgery — during laparoscopy Any adhesions will be noticed, the prevalence of adhesions will be calculated regarding the age, parity, previous history of miscarriage and past medical history.
  The prevalence of adhesions will be calculated according to the indication of laparoscopy.
  The prevalence of adhesions will be compared according to different items. Comparison between patients with no past surgical history and those who have past surgical history.
  Comparison between patients who have history of ectopic pregnancy and those who have no history of ectopic pregnancy.
  Comparison between patients with previous caesarean section and patients with previous other abdominopelvic surgery.

SUMMARY:
To assess the prevalence of surgical adhesions among women undergoing laparoscopy, and the severity of the adhesions according to proposed classification of intra-abdominal adhesions.

DETAILED DESCRIPTION:
Patients will be recruited from the women at Women's Health Hospital Assuit University that will undergo laparoscopy for any cause. After the patients has been examined and put on a list for laparoscopy, they will be counselled about our study and its benefits. Written consent will be obtained.

All women will be subjected to the following:

1. History taking:

   1. Personal history: demographic factors and age.
   2. Obstetric history: parity, last delivery, history of abortion.
   3. Menstrual history: regular or irregular cycles, P/C.
   4. Past history: history of chronic diseases such as diabetes or hypertension, endometriosis, chronic pelvic pain and PID.
   5. Surgical history: of any previous operations including abdomino-pelvic surgery (either laparoscopy or laparotomy) and caesarean section.
   6. The complain of the patient and the indication of laparoscopy.
2. Clinical examination:

   * General examination including pulse, blood pressure, temperature, BMI and pallor.
   * Abdominal examination for scars of previous operations or fundal level.
3. Investigations:

   * Ultrasonography: to assess the uterus and adnexa.
   * Blood sample: it will be examined for the following; complete blood picture and renal function test.
4. During laparoscopy:

   Any adhesions will be noticed, the prevalence of adhesions will be calculated regarding the age, parity, previous history of miscarriage and past medical history.

   The prevalence of adhesions will be calculated according to the indication of laparoscopy.

   The prevalence of adhesions will be compared according to different items. Comparison between patients with no past surgical history and those who have past surgical history.

   Comparison between patients who have history of ectopic pregnancy and those who have no history of ectopic pregnancy.

   Comparison between patients with previous caesarean section and patients with previous other abdominopelvic surgery.
5. The adhesions will be noticed, its site will be detected (between uterus and bladder, uterus and abd. Fascia, uterus and omentum, omentum and abd. Fascia or adhesions to other pelvic structure that interfere with the delivery), its consistency (Filmy or dense) and thickness (either < 3cm, 3-6cm, or > 6cm) and these informations will be subjected to the proposed classification and every case will have its score. The data will be analysed to find out which cases have high score and their common risk factors that are expected to be the cause of this high score.

ELIGIBILITY:
Inclusion Criteria:

* Women who will undergo laparoscopic surgery at Women's Health hospital Assuit University.

women aged 18 years or more.

Exclusion Criteria:

* Women who refused to participate in our study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the women at Women's Health Hospital Assuit University that will undergo laparoscopy for any cause
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of surgical adhesions among women undergoing laparoscopic surgery at Women's Health Hospital (prospective cross-sectional study). | baseline
  the prevalence of surgical adhesions among women undergoing laparoscopy in Women's Health Hospital Assuit University.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut University, Asyut
  - Women's Health Hospital, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboshama RA, Taha OT, Abdel Halim HW, Elrehim EIA, Kamal SHM, ElSherbiny AM, Magdy HA, Albayadi E, Elsaid RE, Abdelghany AM, Anan MA, Abdelfattah LE. Prevalence and risk factor of postoperative adhesions following repeated cesarean section: A prospective cohort study. Int J Gynaecol Obstet. 2023 Apr;161(1):234-240. doi: 10.1002/ijgo.14498. Epub 2022 Oct 26. PMID 36200671